CLINICAL TRIAL: NCT03388671
Title: Laparoscopic Guided Transversus Abdominis Plane Block for Postoperative Analgesia After Pediatric Laparoscopic Surgery.
Acronym: TAB
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300080
Record Dates: First submitted 2017-12-25; First posted 2018-01-03 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dental Occlusion; Bupivacaine; bucain

STUDY DESIGN:
Intervention Model Description: The aim of this study will be to investigate the safety and analgesic efficacy of Transversus Abdominis Plane (TAB) Block versus psoas blocks. Both blocks will be administered surgically and guided by the laparoscopy screen in children undergoing laparoscopic surgery.
Who Masked: Participant, Outcomes Assessor
Masking Description: The data collection personnel and the patients' guardians will be blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAB Block (Active Comparator): Patients will recieve 0.3ml/kg bupivacaine 0.25% on each side for laparoscopically guided Transversus abdominis plane block.
  Interventions: Procedure: TAB Block; Drug: Bupivacaine
- Psoas Block (Active Comparator): Patients will recieve 0.3ml/kg bupivacaine 0.25% on each side for laparoscopically guided psoas block.
  Interventions: Procedure: Psoas Block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: TAB Block — patients will recieve 0.3ml/kg bupivacaine 0.25% on each side for laparoscopically guided TAB Block
  Arms: TAB Block
Procedure: Psoas Block — patients will recieve 0.3ml/kg bupivacaine 0.25% on each side for laparoscopically guided Psoas Block
  Arms: Psoas Block
Drug: Bupivacaine — patients will recieve 0.3ml/kg bupivacaine 0.25% on each side for laparoscopically guided Psoas Block or TAB block
  Other Names: Bucain

SUMMARY:
The aim of this study will be to investigate the safety and analgesic efficacy of Transversus Abdominis Plane (TAB) Block versus psoas block blockade. Both blocks will be administered surgically and guided by the laparoscopy screen in children undergoing laparoscopic surgery.

DETAILED DESCRIPTION:
Transversus abdominis plane (TAP) block is a promising effective method for postoperative pain control after major abdominal surgery. TAP block provides analgesia by inhibiting nerve conduction from the anterior abdominal wall arising from the intercostal nerves, subcostal nerves, and first lumbar nerve (T6-L1). Using a landmark technique, it is easily performed, but its popularity has decreased because of reduced efficacy due to inaccurate injection and the potential for intra-peritoneal organ damage. Ultrasound-guided TAP block provides better results and fewer complications, but it requires experienced operators. Surgically administered TAP (sTAP) block guided by the video camera of the laparoscope is a simple technique and may cause no complications. Also, under laparoscopic guidance, block of ilioinguinal, iliohypogastric, and genitofemoral nerves can be possible with anesthetic injection in the plane between psoas major and the fasciae covering its anterior aspects [laparoscopic-assisted psoas (LAP) blockade].

ELIGIBILITY:
Inclusion Criteria:

* Children (1-6 years) of both sexes undergoing elective laparoscopic surgeries that last >30minutes (eg. undescended testis and inguinal hernia repair).
* Written consent, free and informed

Exclusion Criteria:

* Significant respiratory, cardiac or renal disease
* BMI >95th percentile for age.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2017-12-25 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
FLACC PAIN score | 36hours
  postoperative FLACC pain scores.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdelghaffar, MD, Principal Investigator — Professor in anesthesia and intensive care department, faculty of medicine, Assiut university, Egypt.
Locations (1):
- Pediatric hospital, faculty of medicine, Assiut university, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No